CLINICAL TRIAL: NCT05221281
Title: Implementing a Multimodal RCT Intervention to Improve the Transition of Patients With Crohn's Disease From Pediatric to Adult Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Crohn's and Colitis Canada (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other); The Canadian Children Inflammatory Bowel Disease Network: A Partnership with the CH.I.L.D. Foundation (Unknown); The CH.I.L.D. Foundation - Children with Intestinal & Liver Disorders (Unknown)
Responsible Party: Principal Investigator, Eric Benchimol, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1000078476
Record Dates: First submitted 2022-01-10; First posted 2022-02-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Adolescent Development; Transition; Mental Health Wellness 1
Keywords: Transition from Pediatric to Adult Care; Health Services Research; Adolescent Medicine
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Multimodal intervention consisting of four core components. (Experimental): Core Component 1: Individualized Assessment
  Core Component 2: Transition Facilitation with a Navigator
  Core Component 3: Participant Skills-building
  Core Component 4: Structured Educational eLearning Curriculum
  Interventions: Behavioral: Multimodal intervention consisting of four core components
- Control: Standard of care (Other): Routine Care
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Multimodal intervention consisting of four core components — Core Component 1: Individualized Assessment: Each participant will undergo individualized assessment of their biopsychosocial risk profile (PIBD INTERMED), self-efficacy (IBD-SES-A), function (IBD-DI), transition readiness (TRAQ) and IBD knowledge (IBD-KID2), and depression, anxiety and activation.
  Core Component 2: Transition Navigator: Participants will be assigned a transition navigators, who will have knowledge of IBD, an understanding of the care pathway involved in transitioning IBD patients, and the skills and ability to provide psychosocial support.
  Core Component 3: Participant Skills-building: Skills-building materials delivered virtually. Navigators will also be trained as motivational coaches and will lead separate personalized virtual sessions targeting individual skills that have been identified as deficient during the assessment phase.
  Core Component 4: eLearning Curriculum: Organized online eLearning modules with reinforcement of knowledge by the navigators.
  Arms: Intervention: Multimodal intervention consisting of four core components.
Behavioral: Standard of care — The control group will be provided a standardized version of routine care for transition. In addition to recruiting centers' standard of care, all participating centers will implement the following transition interventions:
  1. A written letter explaining the goals of transition to the patient and family.
  2. Completion of age-appropriate checklists to ensure adolescents are meeting milestones of transition (developed by the TRACC Network).51
  3. Annual online live educational webinars on transition and adolescent issues (hosted by the CIDsCaNN Education Committee).
  4. Completion of the Pediatric INTERMED,52 with appropriate biopsychosocial intervention.
  5. Completion of a transfer-of-care summary letter sent to the receiving adult gastroenterologist using a standardized letter template.53
  The Control Group may also receive any interventions currently in place in their participating care center, but will not receive the formal 4-component intervention described below.
  Other Names: Control
  Arms: Control: Standard of care

SUMMARY:
Background: Transition in care is defined as the "purposeful and planned movement of adolescents and young adults with a chronic medical condition from pediatric to adult-oriented healthcare systems/care providers." Currently, there is no Level 1 evidence of an intervention to improve the care of transitioning adolescents and young adults (AYAs) with inflammatory bowel disease (IBD). The development of a transition program using a biopsychosocial approach will improve the standards for healthcare delivery to transitioning IBD patients. This is a protocol for a structured randomized controlled trial (RCT) to assess the efficacy and impact of a multimodal intervention focused on improving patient function, transition readiness and outcomes among AYA patients with IBD being cared for at pediatric centers in Canada.

Methods: This multi-center RCT is a type 1 hybrid effectiveness-implementation trial to evaluate effectiveness of the intervention and how it can be implemented more widely after the trial. We will include patients aged 16.0 to 17.5 years. The intervention program consists of 4 core components: 1) individualized assessment, 2) transition navigator, 3) virtual patient skills-building with a focus on building resilience, self-management and self-efficacy, and 4) a virtual structured education program. The control group will undergo standard-of-care defined by each participating center. The primary outcome will be the IBD Disability Index, a validated measure to assess patient functioning. Secondary outcomes include transition readiness, anxiety and depression scales, and health service utilization rates. Additionally, we will identify the effectiveness of an evidence-based implementation approach and related barriers and facilitators for the intervention program.

Discussion: The type 1 hybrid effectiveness-implementation design will allow us to develop a feasible, sustainable, and acceptable final intervention model. The intervention will consist of modules that can be accessed in an online, virtual platform. The implementation will not depend on individual hospital resources, allowing centralization of interventions and funding. The authors anticipate that the main study limitation will relate to study subjects not completely adhering to every component of the intervention, which will be evaluated and addressed using the implementation science approach.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-17.5 years
* Diagnosed with IBD diagnosed using standard criteria
* Ability to speak/read English at a functional (Grade 8) level
* Intention to reside in Canada after transfer to adult care
* Ability to use a smartphone or personal computer for the virtual intervention

Exclusion Criteria:

* Do not speak English fluently
* Intention to leave Canada after graduation from high school

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
IBD Disability Index (IBD-DI) | 3 years
  Ordinal variable that measures participant functioning as the primary outcome. IBD-DI was selected as a validated measure of overall disability, functioning, and health. The primary outcome will be measured 3 years after enrollment.

SECONDARY OUTCOMES:
Transition Readiness Assessment Questionnaire (TRAQ) | 3 years
  Transition Readiness
Transition Readiness Assessment Questionnaire (TRAQ) | Up to 24 months (at time of transfer to adult care)
  Transition Readiness
Transition Success Scores (TSS) | 3 years
  Transition Readiness
Transition Success Scores (TSS) | Up to 24 months (at time of transfer to adult care)
  Transition Readiness
Pediatric IBD INTERMED | 3 years
  Biopsychosocial Risk Profile
Pediatric IBD INTERMED | Up to 24 months (at time of transfer to adult care)
  Biopsychosocial Risk Profile
IBD-KID2 | 3 years
  Disease-related knowledge
IBD-KID2 | Up to 24 months (at time of transfer to adult care)
  Disease-related knowledge
IBDQ-32 | 3 years
  Quality of life
IBDQ-32 | Up to 24 months (at time of transfer to adult care)
  Quality of life
IBD Self-Efficacy Scale - Adolescent (IBD-SES-A) | 3 years
  Self-Efficacy
IBD Self-Efficacy Scale - Adolescent (IBD-SES-A) | Up to 24 months (at time of transfer to adult care)
  Self-Efficacy
Physician Global Assessment (PGA) | 3 years
  Physician assessment of disease activity
Physician Global Assessment (PGA) | Up to 24 months (at time of transfer to adult care)
  Physician assessment of disease activity
Fecal calprotectin | 3 years
  Measure of gut inflammation
Modified Harvey-Bradshaw Index (HBI) for Crohn's disease | 3 years
  Disease activity in Crohn's disease patients
Modified Harvey-Bradshaw Index (HBI) for Crohn's disease | Up to 24 months (at time of transfer to adult care)
  Disease activity in Crohn's disease patients
Pediatric Ulcerative Colitis Activity Index (PUCAI) | 3 years
  Disease activity in ulcerative colitis patients
Pediatric Ulcerative Colitis Activity Index (PUCAI) | Up to 24 months (at time of transfer to adult care)
  Disease activity in ulcerative colitis patients
Emergency department visit after 18th birthday (yes/no) | 3 years
  Health services utilization
Number of emergency department visits after 18th birthday | 3 years
  Health services utilization
Hospitalization after 18th birthday (yes/no) | 3 years
  Health services utilization
Number of outpatient visits to a gastroenterologist after 18th birthday | 3 years
  Health services utilization
IBD Disability Index (IBD-DI) | Up to 24 months (at time of transfer to adult care)
  Ordinal variable that measures participant functioning as the primary outcome. IBD-DI was selected as a validated measure of overall disability, functioning, and health.

CONTACTS AND LOCATIONS:
Overall Officials: Eric I Benchimol, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
* Location of the repository - OSF.io or journal (planned)
  * Administrators for the repository Since we are not sure which journals we will submit to at this time, we cannot comment on the location/administrators for the repository.
  * De-identified study data plans - At a minimum, research journals are asking that authors share a 'minimal data set' for submission. This is normally defined as the minimal data set to consist of the data required to replicate all study findings reported in the article, as well as related metadata and methods. This is what will be shared with journals upon submission.
  * Privacy protections for stored study data - Only de-identified study data will be shared with the open access repository. Submission to research journals has been outlined on the participant consent form.

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077
- [Derived] Bollegala N, Barwick M, Fu N, Griffiths AM, Keefer L, Kohut SA, Kroeker KI, Lawrence S, Lee K, Mack DR, Walters TD, de Guzman J, Tersigni C, Miatello A, Benchimol EI. Multimodal intervention to improve the transition of patients with inflammatory bowel disease from pediatric to adult care: protocol for a randomized controlled trial. BMC Gastroenterol. 2022 May 18;22(1):251. doi: 10.1186/s12876-022-02307-9. PMID 35585484